CLINICAL TRIAL: NCT06279858
Title: Probiotic Intervention for Microbiome Modifications and Consequential Clinical Improvements in Children With Fragile X Syndrome: Pilot Study
Brief Title: Probiotic Intervention for Microbiome Modifications and Clinical Improvements in Fragile X Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Specila hospital for cerebral palsy and developmental neurology (Other)
Collaborators: FRAXA Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1-2024
Record Dates: First submitted 2024-02-11; First posted 2024-02-28 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Fragile X Syndrome
Keywords: Fragile X Sindrome; Gut-Brain Axis; Probiotics
MeSH Terms: conditions — Fragile X Syndrome | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: This is open label trial without masking, where each participant receives probiotic for 3 months (12 weeks). It will be single group assignment. In this approach, participants act as their own controls by measuring the microbiome and other parameters before and after taking the probiotics. This design was chosen because individual's microbiome is highly personalized. Even within a family, individuals can have distinct microbiomes. The unique composition of an individual's microbiome can have implications for the effectiveness of probiotics. Thus, changes in analyses and scores between baseline and 3-month study period will be assessed for everyone. Specifically, microbiome modifications that may be associated with changes in behavior and brain processing will be examined.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Probiotics (Experimental): Each participant receives probiotic for 3 months (12 weeks). Participants act as their own controls by measuring the microbiome and other parameters before and after taking the probiotics. This was chosen because individual's microbiome is highly personalized. The unique composition of an individual's microbiome can have implications for the effectiveness of probiotics. All participants will receive probiotic mixture which contains: (i) Lactobacillus casei BL 2401 (40%), (ii) Lactobacillus salivarius BL 2201 (40%) (iii) Bifidobacterium breve BL 3406 (20%). Total amount is 5 x109 CFU in one HPMC capsule, at the end of the shelf life. These strains are registered and preserved in the French National Collection of Cultures of Microorganisms (CNCM, Collection Nationale de Cultures de Microorganismes). They are on EFSA's QPS (Qualified and Presumption of Safety) list and are considered safe for use in food and dietary products
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — Patients will be recruited and included in the study. At baseline, a detailed medical history, and physical and neurological examination will be carried out, with all medications and medical problems documented for all participants. In the first 4 weeks, each patient will receive a weekly call to evaluate tolerability of the probiotic and any adverse events (AEs). Visit 2 will be organized after 6 weeks and final visit 3 after 12 weeks of study period. Any change in medications will also be documented during visits. The examination and documentation of AEs, will be repeated at each visit, while CGI-I will be scoring at visit 2 and final visit 3. Outcome measures will be repeated at the final followup visit at 3 months/end of treatment. Stool samples will be collected twice, at the baseline and final visits. Analyses of microbiome will be performed once, at the end of the study, when all samples are collected and sent to the selected laboratory.

SUMMARY:
The primary objective of this clinical trial is to evaluate efficacy of probiotic mixture which contains Lactobacillus casei, Lactobacillus salivarius and Bifidobacterium breve, in children with Fragile X aged 3-18 years. Specifically, links between microbiome modifications by probiotic mixture and behavioral manifestations and brain processing (eye tracker, EEG analysis) will be assessed. Exploratory objects of this trial are analyses of microbiome composition and assessment of its alterations and modifications (by probiotic mixture) that may lead to clinical improvement and prediction which patients with FXS may be likely to benefit from probiotics treatment.

This is open label trial without masking, where each participant receives probiotic for 3 months (12 weeks). It will be single group assignment. The study plans to enroll 15 participants with FXS, aged 3-18 years, both sexes, during 1-year period and complete all study-related activities by January 2025. During the 3-month study period, subjects will attend three visits (screening/baseline, 6-week, and 3-month visits) to the Fragile X Clinic at the Special Hospital for Cerebral Palsy and Developmental Neurology, Belgrade, Serbia. The primary outcome measureswill be Vineland Adaptive Behavior Scales-Third Edition (VABS-III) and eye tracking measures (social gaze and pupillometry). Exploratory endpoint will be microbiome analyses. Secondary outcome measures will be: CGI-S and CGI-I scores, ABC-CFX score, quality of life, sleep habits and EEG analyses.

DETAILED DESCRIPTION:
One of the initial indicators of health, reflecting an individual's lifestyle and behavioral tendencies, is the human gut microbiome and microbiota. Most of the microbiome development in early human life, along with significant shifts in its composition, occur within the initial 2 to 3 years of existence. Despite ongoing study, a comprehensive comprehension of gut microbiota functionality is yet to be achieved, and its potential impact on various aspects of health and disease remains a complex scientific puzzle. An increasing body of research is focusing on the intricate interplay between the gut microbiome and the central nervous system (CNS). The bidirectional biochemical signaling pathway connecting the gastrointestinal tract and CNS is referred to as the gut-brain axis. This concept has recently been expanded to encompass the "microbiota-gut-brain axis" or MGB axis, highlighting the involvement ofgut microbiota in the biochemical interactions between these two systems. From the moment of birth, chemicals released by the gut microbiota play a pivotal role in shaping brain development. Any disruption in this dynamic interaction significantly heightens the potential for neurodevelopmental disorders (NDDs). Additionally, emerging data indicate that early microbial colonization of the intestinal tract plays a role in regulating neurogenesis in the hippocampus. Moreover, in the context of myelination, a study from Ireland illuminates the potential involvement of the host's microbiota in controlling prefrontal cortex myelination in ice. Germ-free mice exhibit an increased number of hypermyelinated axons, accompanied by pronounced upregulation of genes associated with myelination and myelin flexibility. Lastly, the metabolites produced by the gut microbiota appear to play a role in maintaining the integrity of the host's blood-brain barrier and influencing paracellular permeability. Insights from studies on mouse models provide indications that specific metabolites, such as acetate, propionate, and sodium butyrate, are linked to adjustments in blood-brain barrier integrity. They propose that probiotics could potentially rebalance the microbial composition in the human intestine, thereby playing a role in therapy and prevention of mental health issues like stress and anxiety disorders. Wang et al.'s study of probiotic-prebiotic effects in children diagnosed with autism spectrum disorder (ASD) revealed a reduction in pathogenic bacteria (Clostridium) and an increase in beneficial ones (such as Bifidobacteriales), resulting in decreased ASD severity and gastrointestinal symptoms. This bidirectional communication axis, involving various signaling pathways, presents a vast realm for further exploration. Interventions aimed at modulating the gut microbiota, such as the utilization of antibiotics, probiotics, prebiotics, and potentially fecal microbiota transplantation (FMT), could potentially exert influence over the clinical attributes and progression of NDDs. The most common types of probiotics include Saccharomyces boulardii yeast, as well as species from the Lactobacillus and Bifidobacterium groups. In clinical trials, probiotics showed potential in treating ASD-like behavioral phenotypes and GI symptoms as well as sensory profiles in children with ASDs. In an Egyptian study conducted in an open-label manner, 30 children with autism were given probiotic supplements for a period of three months. Following the supplementation, analysis of stool samples using polymerase chain reaction (PCR) revealed an increase in the population of beneficial bacteria, specifically Lactobacilli and Bifidobacteria. Moreover, noteworthy improvements were observed in the severity of autism symptoms among the participants. This study suggests that probiotic intervention could hold promise as a complementary method to enhance the well-being of individuals with ASD. The observed positive effects on microbial balance and symptom severity point towards a potential avenue for exploring the role of probiotics in augmenting treatment strategies for autism. Probiotics and Gut microbiome in fragile X syndrome (FXS). The role of the gut microbiome in fragile X syndrome (FXS) remains largely unexplored. To our knowledge, the relationship between FXS in humans and gut microbiota has not yet been assessed. However, data obtained from the Fragile X Online Registry with Accessible Database (FORWARD) study revealed that consumption of soy-based infant formula is associated with increased prevalence of autism, GI problems, allergies, and more severe autistic behaviors related to language and self-injurious behavior in individuals with FXS. It should be noted that GI problems were the most frequent reason cited for switching to soy-based infant formula with a 25% reported usage rate in the FORWARD study population, which is significantly higher than the general population. One of possible mechanism underlying soy-induced effects in ASD and FXS could include an altered gut microbiome. In addition, there are several preclinical research which emphasize the role of dysbiosis and/or probiotics in FXS animal models. The mouse and human microbiota share 89% similarity in overall bacterial genera meaning the outcome should be realistic and transferable between species when modeling human disease in animal models. FXS is a prominent example of epigenetic dysregulation and constitutes the most prevalent monogenic cause of and intellectual disability (ID) and autism spectrum disorder (ASD). The syndrome emerges from an elongated CGG trinucleotide repeat expansion exceeding 200 repeats, which leads to transcriptional inhibition due to hypermethylation of the promoter and the repeat region within the 5'-UTR of the fragile X messenger ribonucleoprotein 1 (FMR1) gene. The resultant absence or diminished expression of the encoded gene product, FMRP, underpins the manifestation of FXS. The epigenetic silencing of FMR1, mediated by DNA methylation and histone modifications that lead to FMRP loss, extends its influence across the genome, affecting various non-coding RNAs. Consequently, this disruption impacts the transcription of multiple genes pivotal to synaptic plasticity and neuronal functions, thus contributing to the FXS phenotype. The study conducted in 2022 compared of the epigenetic profiles of two distinct groups of mice: one group that was exposed to Lactobacillus reuteri during their prenatal development, and another group that received a placebo treatment. The investigation focused on 23 specific genes known for their involvement in neurological functions. Notably, a substantial and statistically significant disparity in methylation patterns was identified between these two groups. It is important to acknowledge that the observed differences in methylation might potentially be influenced by genetic variations inherent in the mouse model. Despite this possibility, these findings gain credibility from the significant disparities detected between the control and experimental groups, which included randomly assorted litter mates. Consequently, the researchers were inclined to attribute these findings to the influence of an altered gut microbiota, as suggested by their results.

2. Study Timelines The study plans to enroll 15 participants with FXS, aged 3-18 y. both sexes, during 1-year period and complete all study-related activities by January 2025. During the 3-month study period, subjects will attend three visits to the Special Hospital for Cerebral Palsy and Developmental Neurology, Belgrade, screening/baseline, 6-week, and 3-month visits. In addition, routine phone calls will be made once per week during the first month of the study. This trial has a single-site design. All results and data will be de-identified to protect the confidentiality of the research subject.

3.Objectives Primary objective

1. To evaluate efficacy of probiotic mixture which contains Lactobacillus casei, Lactobacillus salivarius and Bifidobacterium breve, administered orally, once daily, for 12 weeks to children with fragile X syndrome (FXS) aged 3-18 y. on their behavior and brain processing.

   Secondary objectives
2. Assessment of link between: (i) microbiome modifications by probiotic mixture which contains Lactobacillus casei, Lactobacillus salivarius and Bifidobacterium breve, administered orally, once daily, for 12 weeks and (ii) behavioral manifestations in children aged 3 to 18 years diagnosed with FXS.
3. Assessment of link between: (i) microbiome modifications by probiotic mixture which contains Lactobacillus casei, Lactobacillus salivarius and Bifidobacterium breve, administered orally, once daily, for 12 weeks and ii) brain processing (a. event related potential habituation paradigm and social gaze monitoring using the Eye Tracker; b. EEG analysis) in children aged 3 to 18 years diagnosed with FXS.

   Expiratory objective 1. Analyses of microbiome composition and assessment of its alterations and modifications (by probiotic mixture which contains Lactobacillus casei, Lactobacillus salivarius and Bifidobacterium breve, administered orally, once daily, for 12 weeks) that may lead to clinic 4.Hypothesis: Daily intervention with probiotic mixture which contains Lactobacillus casei, Lactobacillus salivarius and Bifidobacterium breve will lead to: (i) significant microbiome modifications (increased diversity of gut microbiota and changes in gut microbiota composition in the direction of beneficial bacteria) and (ii) consequently to clinical improvement in children, both sexes, aged 3 to 18 years diagnosed with FXS during a 3-month treatment period.
4. Hypothesis: Daily intervention with probiotic mixture which contains Lactobacillus casei, Lactobacillus salivarius and Bifidobacterium breve will lead to: (i) significant microbiome modifications (increased diversity of gut microbiota and changes in gut microbiota composition in the direction of beneficial bacteria) and (ii) consequently to clinical improvement in children, both sexes, aged 3 to 18 years diagnosed with FXS during a 3-month treatment period.
5. Study design. This is open label trial without masking, where each participant receives probiotic for 3 months (12 weeks). It will be single group assignment. In this approach, participants act as their own controls by measuring the microbiome and other parameters before and after taking the probiotics. This design was chosen because individual's microbiome is highly personalized. Even within a family, individuals can have distinct microbiomes. The unique composition of an individual's microbiome can have implications for the effectiveness of probiotics. Thus, changes in analyses and scores between baseline and 3-month study period will be assessed for everyone. Specifically, microbiome modifications that may be associated with changes in behavior and brain processing will be examined. The study will be approved by hospital IRB.

Patients (up to 15 individuals aged 3-18 years, both sexes) will be recruited and included in the study within Fragile X Clinic at the Special Hospital for Cerebral Palsy and Developmental Neurology in Belgrade, Serbia (more info at: https://fragilex.org/our-research/fragile-x-clinics/international-support-clinics/#serbia). At baseline, a detailed medical history, and physical and neurological examination will be carried out, with all medications and medical problems documented for all participants. In the first 4 weeks, each patient will receive a weekly call to evaluate tolerability of the probiotic and any adverse events (AEs). Visit 2 will be organized after 6 weeks and final visit 3 after 12 weeks of study period. Any change in medications will also be documented during visits. The examination and documentation of AEs, will be repeated at each visit, while CGI-I will be scoring at visit 2 and final visit 3. Outcome measures will be repeated at the final followup visit at 3 months/end of treatment. Stool samples will be collected twice, at the baseline and final visits. Analyses of microbiome will be performed once, at the end of the study, when all samples are collected and sent to the selected laboratory. The complete schedule of all study procedures is also listed in a table format below. Selected probiotics. All participants will receive probiotic mixture which contains: (i) Lactobacillus casei BL 2401 (40%), (ii) Lactobacillus salivarius BL 2201 (40%) (iii) Bifidobacterium breve BL 3406 (20%). Total amount is 5 x109 CFU in one HPMC capsule, at the end of the shelf life. These strains are registered and preserved in the French National Collection of Cultures of Microorganisms (CNCM, Collection Nationale de Cultures de Microorganismes). They are on EFSA's QPS (Qualified and Presumption of Safety) list and are considered safe for use in food and dietary products. Thanks to its properties, this mixture of strains for human use will act as an aid in the therapy of digestive, skin, respiratory and neurodevelopmental disorders, with the aim of balancing the immune response and restoring the intestinal microbiota and the intestinal barrier. Through genetic mapping, strains were identified according to phenotypic criteria (morphology, biochemical testing, conditions in which they grow) but also according to genotypic criteria (16S rDNA sequencing). In in vitro studies for each of the three specific strains, the following were examined and determined: (i) resistance to conditions in the digestive tract; (ii) adhesion to intestinal mucosa cells; (iii) survivability and long-term stability; (iv) absence of gene transfer for antibiotic resistance; (v) the ability to stimulate the secretion of IL-10 and (vi) antagonism and inhibition of the growth of pathogenic bacteria.

5. Data and Specimen Management and Confidentiality Subjects will be recruited through the Fragile X Clinic at the Special Hospital for Cerebral Palsy and Developmental Neurology, Belgrade, Serbia. Potential subjects who are interested in participating in the study will be pre-screened either via telephone or on site by the research team. This will also allow potential subjects to ask study-related questions and discuss the study in depth with the research team. The review of subjects' medical records is for limited information and only to determine eligibility. The data are derived from clinically indicated procedures and there is minimal risk to the subject. Only research personnel will access medical records. Without an initial review of the medical record for screening purposes, it would not be possible to identify potential subjects and confirm their applicability for study participation. Once eligibility is confirmed, subjects will be approached to obtain their authorization to access and use their health information for the research.Each participant's study records will be filed in a research chart, and subject information will be coded to protect confidentiality. All charts will be kept in a locked cabinet or a locked file room. The identifiers used to identify subjects will be kept in locked offices and/or locked cabinets, and the electronic database containing personal information will be kept on a secure computer network accessible only to PI's research team. We will use the REDCap (Research Electronic Data Capture) system for data management. r. The REDCap system consists of secure, web-based applications that are flexible enough to be used for a variety of types of research, provide an intuitive interface for users to enter data, and have real time validation rules (with automated data type and range checks) at the time of entry. These systems offer easy data manipulation with audit trails for reporting, monitoring, and querying patient records as well as and automated export mechanism to common statistical packages (SPSS, SAS, Stata, R/S-Plus). The subjects' health information, along with the identifiers, will be kept with the investigator, until the conclusion of the study, or when immediate access is no longer required. Thereafter, the information may be transferred to records for long term storage. When the investigator or any regulatory agencies no longer require the information (but no sooner than 5 years), the documents will be securely shredded. All study personnel will have access to study records, data, and specimens. If required, access to study records and data will be made available to representatives of the IRB. Enrolled subjects will be made aware that study personnel, and representatives of the IRB will have access to their records. This will be included in the consent form and will also be thoroughly reviewed during the consent process. All research personnel will have current GCP training for investigators and staff involved in research involving human subjects. In addition, every attempt will be made to ensure that the personal and medical information of the subject will be kept private; however, we cannot guarantee total privacy. The subject's personal and medical information may be given out if required by law. For example, reporting sensitive information (such as child abuse) to local authorities if necessary. The results and data are de-identified to protect patient confidentiality. The analysis of treatment efficacy will be based on changes in analyses and scores between baseline and 3-month study period. The chosen endpoint at 3-month, based on preliminary data, provides a reasonable treatment time period to assess changes in the response and/or correlation between baseline and followup measures.Data Safety and Monitoring Board (DSMB) is not necessary for such research where the effects of probiotic will be examined. Data and/or Specimen Banking Records and documents pertaining to the conduct of this study including Informed Consent Forms, laboratory test results, and medication inventory records, must be retained by the Principal Investigator for at least 5 years after completion or termination of the study, or for the length of time required by relevant national or local health authorities, whichever is longer. After that period of time, the documents may be destroyed, subject to local regulations. Records transferred to another party will be de-identified. Stool samples Banking: All collected samples for microbiome analyses will be de-identified and will only contain the subject's study ID number and date/time of collection. Biological samples will be processed, stored and destroyed in accordance with protocols in place for biological samples.

Withdrawal of Subjects All subjects and their parent/legal authorized guardian will be advised that they are free to withdraw from participation in this study at any time, for any reason, and without prejudice. Every reasonable attempt should be made by the investigator to keep subjects in the study; however, subjects must be withdrawn from the study if they withdraw consent to participate. Investigator must attempt to contact subjects who fail to attend scheduled visits by telephone or other means to exclude the possibility of an AE being the cause of withdrawal. Should this be the cause, the AE must be documented, reported, and followed. The investigator also has the right to withdraw subjects from the study at any time for lack of therapeutic effect that is intolerable or otherwise unacceptable to the subject, for intolerable or unacceptable AEs, inter-current illness, noncompliance with study procedures, administrative reasons, or in the investigator's opinion, to protect the subject's best interest. If a subject is withdrawn before completing the study, the reason for withdrawal and the date of discontinuation will be recorded on the appropriate case report form. Information gathered about a subject who has terminated the study early, as well as any blood and stool samples, will be kept for analysis unless the subject's caregivers specifically ask for this information to be removed from the analysis. Caregivers will be both informed of this as a part of the consent process and also reminded of this in the event of an early termination.

Risks to Subjects The most common anticipated risks due to participation in the study include anxiety, frustration, fatigue, or embarrassment during the answering of questionnaires, study assessments and testing, as well as during he medical history and exam. Breaks will be offered to subjects as needed. Risks associated with blood draws include bruising, soreness, and slight risk of infection at the needle entry site for the blood draw. This site will be carefully cleaned prior to the draw and an appropriate dressing will be applied to the area. Probiotics might cause mild stomach problems, especially the first few days when child starts taking them. Children might have stomach upset, gas, diarrhea. Those symptoms usually go away after body gets used to them.

Weekly phone calls during the first month will be made by study personnel to evaluate the presence of side effects. .

Potential Benefits to Subjects The potential benefits of study participation are that subjects with FXS: 1. may experience an improvement in physical health, behavioral symptoms, and/or cognitive abilities as a result of treatment with probiotic; 2. will undergo neuropsychological assessments, the results of which may be made available to the family of participants on request; 3. will receive medical exams offered through the study. Additionally, a complete blood count will be conducted as a part of this study. Participants will be informed of clinically significant findings from either the medical exam or CBC as appropriate4. will receive microbiome analyses offered through the study. Participants will be informed of clinically significant findings. 5. will understand that they are contributing to the scientific knowledge that may lead to expansion of the targeted treatment options for subjects with FXS.

No other benefits of participation are anticipated.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has Fragile X syndrome with a molecular genetic confirmation of the full FMR1 mutation or mosaicism.
2. Subject is a male or female age 3 to 18 years.
3. Subject must have a parent or caretaker who is willing to participate in the whole study.
4. Subject and caregiver are able to attend the clinic regularly and reliably.
5. Subject and/or subject's parent/legal authorized representative is able to understand, read, write and speak Serbian fluently to complete study-related materials.
6. Behavioral and other non-pharmacological treatments/interventions must be stable for 4 weeks before screening and must remain stable during the period between screening and the commencement of study probiotic, and throughout the study. Minor changes in hours or times of therapy that are not considered clinically significant will not be exclusionary. Changes in therapies provided through a school program, due to school vacations, are allowed.
7. The use of concomitant medications must be stable, in terms of dose and dosing regimen, for at least 4 weeks prior to Screening and must remain stable during the period between Screening and the commencement of the study; every effort should be made to maintain stable regimens of allowed concomitant medications from the time of commencement of double-blind study medication until the last study assessment.
8. Patient's parent(s), legal authorized guardian(s), or consistent caregiver(s) can understand and sign an informed consent form to participate in the study. For subjects who are not their own legal guardian, subject's parent/legal authorized representative is able to understand and sign an informed consent to participate in the study.
9. Subject and/or subject's parent/legal authorized representative is able to understand, read, write, and speak Serbian fluently to complete study-related materials.

Exclusion Criteria:

1. Families that are not cooperative and will not follow through with the demands of this study;
2. Antibiotic use in the last two months (not counting topical antibiotics);
3. Currently taking antibiotics;
4. Any changes in medications, nutritional supplements, therapies, in the last two months, or any plans to change them during the first 3 months of probiotic treatment;
5. Diagnosis of severe gastrointestinal diseases, such as Crohn's Disease, or Ulcerative Colitis;
6. Subject has a life-threatening medical problem or other major systemic illness that compromises health or safety and/or would interfere with this study;
7. Age younger than 3 or older than 18 years.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
1. Vineland Adaptive Behavior Scales-Third Edition (VABS-III) | 3 month
  The Vineland, which is a gold standard test for assessing adaptive behavior that is widely used in clinical trials, will be administered to the parent/caregiver at baseline and end of treatment/week 12. Subtests include Communication, Daily Living Skills, Socialization, Motor Skills, and Adaptive Behavior Composite. The Vineland has been normed for individuals with intellectual disability and ASD. The third edition includes updated item content to streamline similar items and reduce redundancy, to reflect changes in daily living (e.g., technology) and in conceptions of developmental disabilities (e.g., ASD), and to allow for potential cultural differences by using more generalized wording of certain items
Eye tracking | 3 month
  Eye Tracking Measures: Social Gaze and Pupillometry - For individuals with FXS, findings demonstrated that the social gaze measure shows decreased visual fixations on the eye region while viewing human faces (with greater fixation to the nose region), and these individuals show abnormal pupillary dilation, an indication of sympathetic nervous system reactivity, compared with controls [31].
  During the experiment, individuals with FXS will sit in front of the monitor at the distance of 65 cm, while stimuli consist of human faces in natural size with different emotional expressions will be presented. This eyetracking system has several benefits that make it conducive to testing individuals with developmentaldisorders, including 35 cm x 30 cm of tolerance to head-motion at 65 cm distance without requiring any head apparatus or restraints.

SECONDARY OUTCOMES:
Clinical Global Impression Scales of Severity (CGI-S) and Improvement (CGI-I) - | 3 month
  These scales are standard assessment for medication studies because it allows the clinician to utilize the history from the parent or caretaker and incorporate it into a clinical rating for the clinical follow up of the patient through the treatment trial. In the initial evaluation of the patient, we will use the CGI-S (severity) to judge the severity of the symptoms with a scale of normal, not at all ill; borderline ill; mildly ill; moderately ill; markedly ill; severely ill; or among the most extremely ill. The CGI-S scale will be utilized at the baseline, the week 6, and end of treatment/week 12 follow-up visits The CGI-I scale will be utilized at the week 6 and end of treatment/week 12 follow-up visits. We will use CGI-I to look at improvement or worsening of symptoms with a scale of very much improved; much improved; minimal improvement; no improvement; minimally worse; or very much worse
The Aberrant Behavior Checklist - Community Edition (ABC-C), scored using the FXS-specific factoring system (ABC-CFX) | 3 month
  This measure will be completed by the parent/caregiver at baseline, and end of treatment/week 12. This parent/caregiver report measure is the gold standard measure of problem and interfering behaviors in clinical trials in developmental disabilities. The ABC asks responders to rate behaviors from 0 "not a problem at all" to 3 "the problem is severe in degree" across 58 questions. Its use has been validated in a variety of clinical populations, including in ASD and FXS, has been used extensively in clinical trials. It has been subjected to utility analysis in FXS and linked to caregiver stress in families [36, 37]. Scores will be analyzed using the FXS-specific factor structure such that 54 of the items resolve into 6 subscales (irritability, lethargy, social avoidance, stereotypic behavior, hyperactivity, and inappropriate speech).
Pediatric Quality of Life Questionnaire (PedsQL) Parent Proxy | 3 month
  This measure consists of a series of questions relating to a child's quality of life and is administered to the caregiver of the child. The parent proxy module designed for children 8-12 years of age will be administered to the caregivers of all subjects, regardless of age, because the questions therein are most appropriate for the overall study population's cognitive age and ability. It will be completed at baseline, week 6, and end of treatment/week 12. For any subjects not in school, questions pertaining to "school" will be replaced with references to "work" or other activities in their life
Child Sleep Habits Questionnaire (CSHQ) | 3 month
  This measure consists of a series of questions relating to the sleep habits of children. It will be completed by caregivers of all subjects, regardless of age, at baseline, and end of treatment/week 12.
EEG analyses | 3 month
  One outcome measure involves examining EEG differences observed in individuals with FXS, such as amplified N1 ERP amplitudes, heightened resting gamma power, and decreased gamma phase-locking in sensory cortices. These EEG abnormalities are believed to signify cortical hyperexcitability resulting from an imbalance between excitatory (glutamate) and inhibitory (GABAergic) mechanisms in FXS, which has been the focus of numerous pharmaceutical remediation studies. We are analyze power in alpha and delta band.

OTHER OUTCOMES:
Microbiome analyses | 3 month
  Microbiome modification (increased diversity of gut microbiota and changes in gut microbiota composition in the direction of beneficial bacteria) before and after probiotics' treatment will be assessed and linked with potential behavioral changes and changes in brain processing in children with FXS. Briefly, DNA extraction will be performed by using the AllPrep Power Fecal DNA/RNA kit (Qiagen, Hilden, Germany), according to the manufacturer's instructions. Profiling of bacteria will be performed by 16S rRNA gene sequencing, using primers targeting V3-V4 region, as recommended by Angebault et al, 2020 [40].
  Library preparation will include a single PCR step following a dual barcoding approach. Amplicons library will be sequenced using a MiSeq Reagent Kit v3 (600-cycle) on a Miseq plattform (Illumina).
  The generated raw outputs (in fastq format) will be analyzed with dada2 R package [41].

CONTACTS AND LOCATIONS:
Overall Officials: Dragana Protic, Prof, Principal Investigator — University od Belgrade
Locations (1):
- Special Hospital for Cerebral Palsy and Developmental Neurology, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alam S, Westmark CJ, McCullagh EA. Diet in treatment of autism spectrum disorders. Front Neurosci. 2023 Jul 10;16:1031016. doi: 10.3389/fnins.2022.1031016. eCollection 2022. PMID 37492195
- [Background] Ardissone AN, de la Cruz DM, Davis-Richardson AG, Rechcigl KT, Li N, Drew JC, Murgas-Torrazza R, Sharma R, Hudak ML, Triplett EW, Neu J. Meconium microbiome analysis identifies bacteria correlated with premature birth. PLoS One. 2014 Mar 10;9(3):e90784. doi: 10.1371/journal.pone.0090784. eCollection 2014. PMID 24614698
- [Background] Dimitroglou M, Iliodromiti Z, Christou E, Volaki P, Petropoulou C, Sokou R, Boutsikou T, Iacovidou N. Human Breast Milk: The Key Role in the Maturation of Immune, Gastrointestinal and Central Nervous Systems: A Narrative Review. Diagnostics (Basel). 2022 Sep 12;12(9):2208. doi: 10.3390/diagnostics12092208. PMID 36140609
- [Background] Dominguez-Bello MG, Costello EK, Contreras M, Magris M, Hidalgo G, Fierer N, Knight R. Delivery mode shapes the acquisition and structure of the initial microbiota across multiple body habitats in newborns. Proc Natl Acad Sci U S A. 2010 Jun 29;107(26):11971-5. doi: 10.1073/pnas.1002601107. Epub 2010 Jun 21. PMID 20566857
- [Background] Holt PG. Environmental factors and primary T-cell sensitisation to inhalant allergens in infancy: reappraisal of the role of infections and air pollution. Pediatr Allergy Immunol. 1995 Feb;6(1):1-10. doi: 10.1111/j.1399-3038.1995.tb00250.x. No abstract available. PMID 7550758
- [Background] Wang Y, Kasper LH. The role of microbiome in central nervous system disorders. Brain Behav Immun. 2014 May;38:1-12. doi: 10.1016/j.bbi.2013.12.015. Epub 2013 Dec 25. PMID 24370461
- [Background] Sudo N, Chida Y, Aiba Y, Sonoda J, Oyama N, Yu XN, Kubo C, Koga Y. Postnatal microbial colonization programs the hypothalamic-pituitary-adrenal system for stress response in mice. J Physiol. 2004 Jul 1;558(Pt 1):263-75. doi: 10.1113/jphysiol.2004.063388. Epub 2004 May 7. PMID 15133062
- [Background] Cryan JF, O'Riordan KJ, Cowan CSM, Sandhu KV, Bastiaanssen TFS, Boehme M, Codagnone MG, Cussotto S, Fulling C, Golubeva AV, Guzzetta KE, Jaggar M, Long-Smith CM, Lyte JM, Martin JA, Molinero-Perez A, Moloney G, Morelli E, Morillas E, O'Connor R, Cruz-Pereira JS, Peterson VL, Rea K, Ritz NL, Sherwin E, Spichak S, Teichman EM, van de Wouw M, Ventura-Silva AP, Wallace-Fitzsimons SE, Hyland N, Clarke G, Dinan TG. The Microbiota-Gut-Brain Axis. Physiol Rev. 2019 Oct 1;99(4):1877-2013. doi: 10.1152/physrev.00018.2018. PMID 31460832
- [Background] Carabotti M, Scirocco A, Maselli MA, Severi C. The gut-brain axis: interactions between enteric microbiota, central and enteric nervous systems. Ann Gastroenterol. 2015 Apr-Jun;28(2):203-209. PMID 25830558
- [Background] Dash S, Syed YA, Khan MR. Understanding the Role of the Gut Microbiome in Brain Development and Its Association With Neurodevelopmental Psychiatric Disorders. Front Cell Dev Biol. 2022 Apr 14;10:880544. doi: 10.3389/fcell.2022.880544. eCollection 2022. PMID 35493075
- [Background] Humann J, Mann B, Gao G, Moresco P, Ramahi J, Loh LN, Farr A, Hu Y, Durick-Eder K, Fillon SA, Smeyne RJ, Tuomanen EI. Bacterial Peptidoglycan Traverses the Placenta to Induce Fetal Neuroproliferation and Aberrant Postnatal Behavior. Cell Host Microbe. 2016 Mar 9;19(3):388-99. doi: 10.1016/j.chom.2016.02.009. PMID 26962947
- [Background] Erny D, Hrabe de Angelis AL, Jaitin D, Wieghofer P, Staszewski O, David E, Keren-Shaul H, Mahlakoiv T, Jakobshagen K, Buch T, Schwierzeck V, Utermohlen O, Chun E, Garrett WS, McCoy KD, Diefenbach A, Staeheli P, Stecher B, Amit I, Prinz M. Host microbiota constantly control maturation and function of microglia in the CNS. Nat Neurosci. 2015 Jul;18(7):965-77. doi: 10.1038/nn.4030. Epub 2015 Jun 1. PMID 26030851
- [Background] Hoban AE, Stilling RM, Ryan FJ, Shanahan F, Dinan TG, Claesson MJ, Clarke G, Cryan JF. Regulation of prefrontal cortex myelination by the microbiota. Transl Psychiatry. 2016 Apr 5;6(4):e774. doi: 10.1038/tp.2016.42. PMID 27045844
- [Background] Parker A, Fonseca S, Carding SR. Gut microbes and metabolites as modulators of blood-brain barrier integrity and brain health. Gut Microbes. 2020;11(2):135-157. doi: 10.1080/19490976.2019.1638722. Epub 2019 Aug 1. PMID 31368397
- [Background] Braniste V, Al-Asmakh M, Kowal C, Anuar F, Abbaspour A, Toth M, Korecka A, Bakocevic N, Ng LG, Kundu P, Gulyas B, Halldin C, Hultenby K, Nilsson H, Hebert H, Volpe BT, Diamond B, Pettersson S. The gut microbiota influences blood-brain barrier permeability in mice. Sci Transl Med. 2014 Nov 19;6(263):263ra158. doi: 10.1126/scitranslmed.3009759. PMID 25411471
- [Background] Wang Y, Li N, Yang JJ, Zhao DM, Chen B, Zhang GQ, Chen S, Cao RF, Yu H, Zhao CY, Zhao L, Ge YS, Liu Y, Zhang LH, Hu W, Zhang L, Gai ZT. Probiotics and fructo-oligosaccharide intervention modulate the microbiota-gut brain axis to improve autism spectrum reducing also the hyper-serotonergic state and the dopamine metabolism disorder. Pharmacol Res. 2020 Jul;157:104784. doi: 10.1016/j.phrs.2020.104784. Epub 2020 Apr 17. PMID 32305492
- [Background] Vendrik KEW, Ooijevaar RE, de Jong PRC, Laman JD, van Oosten BW, van Hilten JJ, Ducarmon QR, Keller JJ, Kuijper EJ, Contarino MF. Fecal Microbiota Transplantation in Neurological Disorders. Front Cell Infect Microbiol. 2020 Mar 24;10:98. doi: 10.3389/fcimb.2020.00098. eCollection 2020. PMID 32266160
- [Background] Iliodromiti Z, Triantafyllou AR, Tsaousi M, Pouliakis A, Petropoulou C, Sokou R, Volaki P, Boutsikou T, Iacovidou N. Gut Microbiome and Neurodevelopmental Disorders: A Link Yet to Be Disclosed. Microorganisms. 2023 Feb 15;11(2):487. doi: 10.3390/microorganisms11020487. PMID 36838452
- [Background] Westmark CJ, Kniss C, Sampene E, Wang A, Milunovich A, Elver K, Hessl D, Talboy A, Picker J, Haas-Givler B, Esler A, Gropman AL, Uy R, Erickson C, Velinov M, Tartaglia N, Berry-Kravis EM. Soy-Based Infant Formula is Associated with an Increased Prevalence of Comorbidities in Fragile X Syndrome. Nutrients. 2020 Oct 14;12(10):3136. doi: 10.3390/nu12103136. PMID 33066511
- [Background] Harris SW, Hessl D, Goodlin-Jones B, Ferranti J, Bacalman S, Barbato I, Tassone F, Hagerman PJ, Herman H, Hagerman RJ. Autism profiles of males with fragile X syndrome. Am J Ment Retard. 2008 Nov;113(6):427-38. doi: 10.1352/2008.113:427-438. PMID 19127654
- [Background] Verheij C, Bakker CE, de Graaff E, Keulemans J, Willemsen R, Verkerk AJ, Galjaard H, Reuser AJ, Hoogeveen AT, Oostra BA. Characterization and localization of the FMR-1 gene product associated with fragile X syndrome. Nature. 1993 Jun 24;363(6431):722-4. doi: 10.1038/363722a0. PMID 8515814
- [Background] AlOlaby RR, Zafarullah M, Barboza M, Peng G, Varian BJ, Erdman SE, Lebrilla C, Tassone F. Differential Methylation Profile in Fragile X Syndrome-Prone Offspring Mice after in Utero Exposure to Lactobacillus Reuteri. Genes (Basel). 2022 Jul 22;13(8):1300. doi: 10.3390/genes13081300. PMID 35893036
- [Background] Varian BJ, Weber KT, Kim LJ, Chavarria TE, Carrasco SE, Muthupalani S, Poutahidis T, Zafarullah M, Al Olaby RR, Barboza M, Solakyildirim K, Lebrilla C, Tassone F, Wu F, Alm EJ, Erdman SE. Maternal Microbiota Modulate a Fragile X-like Syndrome in Offspring Mice. Genes (Basel). 2022 Aug 8;13(8):1409. doi: 10.3390/genes13081409. PMID 36011319
- [Background] Farzin F, Rivera SM, Hessl D. Brief report: Visual processing of faces in individuals with fragile X syndrome: an eye tracking study. J Autism Dev Disord. 2009 Jun;39(6):946-52. doi: 10.1007/s10803-009-0744-1. Epub 2009 Apr 28. PMID 19399604
- [Background] Miller LJ, McIntosh DN, McGrath J, Shyu V, Lampe M, Taylor AK, Tassone F, Neitzel K, Stackhouse T, Hagerman RJ. Electrodermal responses to sensory stimuli in individuals with fragile X syndrome: a preliminary report. Am J Med Genet. 1999 Apr 2;83(4):268-79. PMID 10208160
- [Background] Sansone SM, Widaman KF, Hall SS, Reiss AL, Lightbody A, Kaufmann WE, Berry-Kravis E, Lachiewicz A, Brown EC, Hessl D. Psychometric study of the Aberrant Behavior Checklist in Fragile X Syndrome and implications for targeted treatment. J Autism Dev Disord. 2012 Jul;42(7):1377-92. doi: 10.1007/s10803-011-1370-2. PMID 21972117
- [Background] Kerr C, Breheny K, Lloyd A, Brazier J, Bailey DB Jr, Berry-Kravis E, Cohen J, Petrillo J. Developing a utility index for the Aberrant Behavior Checklist (ABC-C) for fragile X syndrome. Qual Life Res. 2015 Feb;24(2):305-14. doi: 10.1007/s11136-014-0759-8. Epub 2014 Jul 26. PMID 25063082
- [Background] Bailey DB Jr, Raspa M, Bishop E, Mitra D, Martin S, Wheeler A, Sacco P. Health and economic consequences of fragile X syndrome for caregivers. J Dev Behav Pediatr. 2012 Nov-Dec;33(9):705-12. doi: 10.1097/DBP.0b013e318272dcbc. PMID 23117595
- [Background] Fitzpatrick SE, Schmitt LM, Adams R, Pedapati EV, Wink LK, Shaffer RC, Sage J, Weber JD, Dominick KC, Erickson CA. Pediatric Quality of Life Inventory (PedsQL) in Fragile X Syndrome. J Autism Dev Disord. 2020 Mar;50(3):1056-1063. doi: 10.1007/s10803-019-04292-7. PMID 31728808
- [Background] Kenny A, Wright D, Stanfield AC. EEG as a translational biomarker and outcome measure in fragile X syndrome. Transl Psychiatry. 2022 Jan 24;12(1):34. doi: 10.1038/s41398-022-01796-2. PMID 35075104
- [Background] Angebault C, Payen M, Woerther PL, Rodriguez C, Botterel F. Combined bacterial and fungal targeted amplicon sequencing of respiratory samples: Does the DNA extraction method matter? PLoS One. 2020 Apr 28;15(4):e0232215. doi: 10.1371/journal.pone.0232215. eCollection 2020. PMID 32343737
- [Background] Belheouane M, Hermes BM, Van Beek N, Benoit S, Bernard P, Drenovska K, Gerdes S, Glaser R, Goebeler M, Gunther C, von Georg A, Hammers CM, Holtsche MM, Homey B, Horvath ON, Hubner F, Linnemann B, Joly P, Marton D, Patsatsi A, Pfohler C, Sardy M, Huilaja L, Vassileva S, Zillikens D, Ibrahim S, Sadik CD, Schmidt E, Baines JF. Characterization of the skin microbiota in bullous pemphigoid patients and controls reveals novel microbial indicators of disease. J Adv Res. 2023 Feb;44:71-79. doi: 10.1016/j.jare.2022.03.019. Epub 2022 Apr 4. PMID 35581140